CLINICAL TRIAL: NCT02017522
Title: Non-Invasive Characterization in Cardiac Sarcoidosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor initial results. Scans were of insufficient quality for study purpose.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Venkatesh L. Murthy, M.D., Ph.D., Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00079881
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Cardiac Sarcoidosis
Keywords: PET; Cardiac sarcoidosis; FDG; Cardiac MRI

STUDY DESIGN:
Intervention Model Description: Subjects will have be injected 11C-PBR28, a compound used as a radiotracer. They will then have a PET CT scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- 11C-PBR PET (Experimental): Subjects will have a blood sample drawn to evaluate the presence of a specific genetic variation which would prevent the new type of imaging test we are evaluating from working and we will test the inflammatory cells in the blood for the same purpose.
  All participants who proceed will have to return on at least one additional day to undergo a positron emission tomography (PET) scan similar to the scan your doctor ordered. we will use 11C-PBR28 as the radiotracer. This study will evaluate whether 11C-PBR28 can show areas of inflammation due to cardiac sarcoidosis. On either the same day or a different day, you will also undergo a cardiac MRI.
  Interventions: Device: 11C-PBR PET

INTERVENTIONS:
Device: 11C-PBR PET — Subjects will have a positron emission tomography (PET) CT scan using 11C-PBR28 as a radiotracer. This study will evaluate inflammation due to cardiac sarcoidosis. The CT scan will improve the images. The total scan time will be about 30 minutes. There will also be some time required for prep, such as inserting an intravenous (IV) catheter in an arm or forearm. Including prep time, the scan will take approximately two hours.
  Subjects will also undergo a cardiac MRI. Cardiac MRI uses strong magnetic fields to make pictures of the heart. We will use gadolinium containing contrast material, given through an intravenous (IV) catheter to highlight areas of scar in your heart which may be due to cardiac sarcoidosis. This scan will take about 60 minutes.

SUMMARY:
In a study of Cardiac sarcoidosis, a serious heart condition, a radiotracer is being used to examine inflammation.

DETAILED DESCRIPTION:
Cardiac sarcoidosis is a serious medical condition which affects the heart. The purpose of this study is to characterize the relationship between the FDG PET findings and other markers of inflammation including using a new targeted PET radiotracer, 11C-PBR28, and analysis of blood specimens.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. must have undergone a cardiac positron emission tomography (PET) scan using 18F-fluorodeoxyglucose (FDG) for clinical reasons (i.e. referred by your doctor) within the preceding 30 days which showed evidence of active inflammation in your heart.

Exclusion Criteria:

1. If you have two copies of a genetic variation called rs6971 which will prevent this tracer from generating high-quality images you may not participate. If you consent, a blood sample will be drawn to check whether you have this genetic variation.
2. Pregnancy or breastfeeding. If you are female and still experience menstrual periods, you must be willing to use contraception until your participation in the study is complete.
3. Allergy or intolerance to contrast dye containing gadolinium
4. Claustrophobia which would prevent you from completing an approximately one hour MRI scan
5. Inability to lie flat with your arms by your head
6. Abnormal kidney function (estimated GFR(glomerular filtration rate) <60 ml/min/1.73 m2)
7. Implanted pacemaker, defibrillator or other medical devices which are not safe for 3 Tesla MRI
8. Metal in the eyes or shrapnel in the body
9. If you are clinically unstable you may not participate in this study. For example, if you have potentially life threatening abnormal heart rhythms which are not controlled by medication or other treatments, you cannot participate. Also, if you need medications to increase your blood pressure or cardiac function due to weak heart muscle, you cannot participate.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-04-04 (Actual); Primary Completion 2015-07-07 (Actual); Study Completion 2015-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh L. Murthy, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five potential participants signed consents, but only three passed screening.
Groups:
- 11C-PBR PET: Subjects will have a blood sample drawn to evaluate the presence of a specific genetic variation which would prevent the new type of imaging test from working.
  All participants who proceed will return on at least one additional day to undergo a positron emission tomography (PET) scan with 11C-PBR28 as the radiotracer to evaluate inflammation due to cardiac sarcoidosis.
Period: Overall Study
Arm/Group | 11C-PBR PET
Started | 3
Scan | 2
Completed | 2
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- 11C-PBR PET: Subjects will have a blood sample drawn to evaluate the presence of a specific genetic variation which would prevent the new type of imaging test we are evaluating from working and we will test the inflammatory cells in the blood for the same purpose.
  All participants who proceed will have to return on at least one additional day to undergo a positron emission tomography (PET) scan similar to the scan your doctor ordered with 11C-PBR28 as the radiotracer. On either the same day or a different day, participants will also undergo a cardiac MRI.
Arm/Group | 11C-PBR PET
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Ratio of 11C-PBR28 in the Myocardium
Description: The primary outcome of this study will be the ratio of 11C-PBR28 PET activity in myocardial regions with inflammation indicated by FDG PET and/or edema indicated by increased T2 signal with cardiac MRI compared to the 11C-PBR28 PET activity in myocardial segments which appear normal on FDG PET and cardiac MRI. The primary outcome is thus the intensity of uptake in abnormal regions as a percentage of the intensity of uptake in normal segments.
Time Frame: 1 hour scan
Population: Insufficient myocardial tissue contrast to define abnormal and normal regions.
Groups:
- 11C-PBR PET: Characters remaining: 623 Subjects will have a blood sample drawn to evaluate the presence of a specific genetic variation which would prevent the new type of imaging test from working.
  All participants who proceed will return on at least one additional day to undergo a positron emission tomography (PET) scan with 11C-PBR28 as the radiotracer to evaluate inflammation due to cardiac sarcoidosis.
Arm/Group | 11C-PBR PET
Number analyzed (Participants) | 0

2. Secondary Outcome: The Ratio of 11C-PBR28 PET Activity in Cardiac Regions With Fibrosis
Description: As a secondary outcome of this study we will evaluate the ratio of 11C-PBR28 PET activity in regions with fibrosis indicated by decreased myocardial perfusion on 82Rb PET and/or late gadolinium enhancement on cardiac MRI without imaging signs of active inflammation compared to 11C-PBR28 PET activity in myocardial segments which appear normal on 82Rb PET, FDG PET and cardiac MRI. This outcome will thus be expressed by 11C-PBR28 PET uptake in fibrotic regions as a percentage of uptake in normal segments
  We will also evaluate the concordance between extracardiac activity seen in 11C-PBR28 and FDG PET, and when available, histopathology of contemporaneous biopsy specimens.
Time Frame: 1 hour scan
Population: Because the two scans performed provided inadequate clarity to allow any analysis, the additional measurements anticipated as secondary were not feasible.
Arm/Group | 11C-PBR PET
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: about 2 hours
Groups:
- 11C-PBR PET: Subjects will have a blood sample drawn to evaluate the presence of a specific genetic variation which would prevent the new type of imaging test being evaluated.
  All participants who proceed will have to return on at least one additional day to undergo a positron emission tomography (PET) scan similar to the scan that their treating doctor ordered. 11C-PBR28 will be used as the radiotracer. On either the same day or a different day, a cardiac MRI will be performed.
Arm/Group | 11C-PBR PET
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No